CLINICAL TRIAL: NCT04334642
Title: Mindfulness and Paralympic Sport: a Mindfulness Based Intervention for Paralympic Boccia Brazilian Team (MPS)
Brief Title: Mindfulness and Paralympic Sport: a Mindfulness Based Intervention for Paralympic Boccia Brazilian Team
Acronym: MPS
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Centro Mente Aberta de Mindfulness (Other)
Responsible Party: Principal Investigator, Marcelo Demarzo, MD, PhD, Head and Associate Professor, Centro Mente Aberta de Mindfulness
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: 19577519.2.0000.5505
Record Dates: First submitted 2020-03-24; First posted 2020-04-06 (Actual); Last update posted 2021-02-10 (Actual); Status verified 2021-02

CONDITIONS: Stress
Keywords: Paralympic Games; Mindfulness; Sport; Athletes; Boccia

STUDY DESIGN:
Intervention Model Description: The research will have as a convenience sample Athletes from the Paralympic Boccia Brazilian Team, which will be compared with itself in the data analysis.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Athletes from the Paralympic Boccia Brazilian Team (Experimental): The research will have as a convenience sample 11 Athletes from the Paralympic Boccia Brazilian Team, which will be compared with itself in the data analysis. This study includes the category called Other participants formed by staff, freshmen, technicians and other professionals who are present during the interventions.
  Interventions: Other: A mindfulness based intervention

INTERVENTIONS:
Other: A mindfulness based intervention — It is a pilot study of feasibility and preliminary effectiveness composed of a longitudinal intervention that uses as a baseline measure a Mindfulness Training of 2 cycles (each cycle is formed by 4 days of intervention); two follow-up measures (1 and 6 months after the 2nd cycle); and a final measurement (12 months after the start of the study).
  Other Names: Mindfulness Training; MBHP

SUMMARY:
The approach of the Tokyo 2020 Paralympic Games brings an opportunity for reflection on how the academic universe follows the evolution of this sports segment and whether it is possible to carry out an intervention that will contribute to improving and maintaining the performance of Paralympic Boccia Brazilian Team. Mindfulness means being aware and describes a natural human capacity that can be trained and previous researches indicate that the presence of mindfulness traits in athletes can be improved with mindfulness training. Specifically, the Paralympic Boccia is a sport that is on the rise for new resources that can collaborate with its performance in a national and international context. Thus, the objective of this study is to evaluate the effects of a mindfulness-based intervention on Paralympic Boccia athletes, in particular, the impact on sports performance and quality of life from the change in attentional level. It is a pilot study of feasibility and preliminary effectiveness composed of a longitudinal intervention that uses as a baseline measure a Mindfulness Training of 2 cycles (each cycle is formed by 4 days of intervention); two follow-up measures (1 and 6 months after the 2nd cycle); and a final measurement (12 months after the start of the study). The research will have as a convenience sample Athletes from the Paralympic Boccia Brazilian Team, which will be compared with itself in the data analysis. It is expected to show a positive impact on the athletes' quality of life (primary outcome). As secondary outcomes, it is expected to show the evolution of sports performance in relation to the accuracy of the pitch and the speed of the ball, in addition to improving the attention focus and perceived stress, which affect the tactics and performance of the game. The potential benefits of this research also have a social component, by expanding the understanding of human nature through sport, and also a functional component, by impacting the performance of these high-performance athletes.

DETAILED DESCRIPTION:
Since the participation of an athlete with a disability in the Olympic Games in 1904, a long road has been traveled until the Paralympic sport was understood as a standard of high performance, in which Brazil stands out when occupying the eighth place in the overall ranking of medals in the Rio 2016 Games, as well as consecutive leader in the Pan American Games (2007, 2011, 2015 and 2019). The approach of the Tokyo 2020 Paralympics brings an opportunity for reflection on how the academic universe follows the evolution of this sports segment and whether it is possible to carry out an intervention that will contribute to improving and maintaining the performance of these athletes.

Mindfulness means being aware and describes a natural human capacity that can be trained. The option of the Paralympic Boccia Brazilian Team for a research on mindfulness is because of the identification of previous researches that indicate that the presence of mindfulness traits in athletes can be improved with mindfulness training. Specifically, the Paralympic Boccia is a sport that is on the rise for new resources that can collaborate with its performance in a national and international context.

Considering that sports performance is composed of several pillars, such as physical, technical, tactical and psychological, there is an opportunity to investigate the following findings of mindfulness-based interventions in a complex population:

Mindfulness practice consistently and significantly improves levels of mindfulness across various sports disciplines.

Physiological and psychological performance improved significantly until the practice of mindfulness.

Based on the available evidence, the practice of mindfulness can be considered as a supplementary training approach to improve performance in precision sports disciplines.

Thus, the objective of this study is to evaluate the effects of a mindfulness-based intervention (MBI) on Paralympic Boccia athletes, in particular, the impact on sports performance and quality of life from the change in attentional level. It is an exploratory study (pilot) to verify if the intervention will be well accepted by the participants (feasibility) and if it will be effective to reproduce the expected effects (preliminary effectiveness) composed of a longitudinal intervention that uses as a baseline measure a Mindfulness Training of 2 cycles (each cycle is formed by 4 days of intervention); two follow-up measures (1 and 6 months after the 2nd cycle); and a final measurement (12 months after the start of the study).

The research will have as a convenience sample 11 Athletes from the Paralympic Boccia Brazilian Team, which will be compared with itself in the data analysis. This study includes the category called "Other participants" formed by staff, freshmen, technicians and other professionals who are present during the interventions. In this way, the participants totalize 25 people: there are eleven athletes categorized as "Athletes" and 14 professionals in the "Other Participants" category. The measure instruments used in the Athletes category will be the same in the Other participants category, with the exception of Performance Evaluation applied only to Athletes.

The methodological procedures of the present work were prepared within the fundamental ethical and scientific procedures, as provided for in Resolution No. 466 of December 12, 2012 of the National Health Council of Ministry of Health, being approved by the Research Ethics Committee (CEP), by protocol 19577519.2.0000.5505.

The intervention will take place at the Brazilian Paralympic Training Center - CTPB, in the City of São Paulo, SP, where an certified instructor with extensive experience in leading groups by Centro Mente Aberta - UNIFESP will conduct the MBI and recommend to athletes to incorporate formal and informal care practices into their daily lives.

It is expected to show a positive impact on the athletes' quality of life (primary outcome). As secondary outcomes, it is expected to show the evolution of sports performance in relation to the accuracy of the pitch and the speed of the ball, in addition to improving the attention focus and perceived stress, which affect the tactics and performance of the game. The potential benefits of this research also have a social component, by expanding the understanding of human nature through sport, and also a functional component, by impacting the performance of these high-performance athletes. In this sense, it produces practical scientific knowledge that can pave the way for the subsequent realization of a large-scale trial that will benefit the greatest number of people.

The investigation is limited by the lack of additional comparison groups and the small sample size to detect effects. However, this is justified by being Paralympic medalists who have a series of unique characteristics, according to the functional classification that includes people with severe or severe motor disabilities, caused basically by cerebral palsy, cervical spinal cord injuries and muscular dystrophies.

The relevance of this research is in its pioneering spirit and originality when evaluating the first intervention based on mindfulness with Paralympic athletes held in Brazil.

ELIGIBILITY:
Inclusion Criteria:

- Must be an Athlete from the Paralympic Boccia Brazilian Team

Exclusion Criteria:

* Diagnosis of an active mental disorder, such as depression and anxiety, in the initial phase of treatment
* Diagnosis of an active mental disorder, such as depression and anxiety, with severe symptoms
* Having previous experience with mindfulness (regular practice in the last 6 months)
* Athletes without access to the internet or electronic means to access audio practices

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2019-06-30 (Actual); Primary Completion 2020-12-10 (Actual); Study Completion 2021-04-25 (Estimated)

PRIMARY OUTCOMES:
Change in quality of life | T0 (baseline), T1 (1 week), T2 (1 month), T3 (6 months), T4 (12 months)
  WHOQOL-bref means World Health Organization Quality of Life Assessment - bref. This Scale assesses quality of life: it is an abbreviated version of the WHOQOL-100 with 26 questions divided into four domains, namely, physical, psychological, social relations and the environment. The answers follow a Likert scale (from 1 to 5, how much the higher the score the better the quality of life).

SECONDARY OUTCOMES:
Change of sports performance | T0 (baseline), T4 (12 months)
  The Pitch Accuracy Test used by the Brazilian Boccia Team in a regular basis.
Change of sports performance (II) | T0 (baseline), T4 (12 months)
  The Ball Speed Test used by the Brazilian Boccia Team in a regular basis.

OTHER OUTCOMES:
Change of attention focus and perceived stress | T0 (baseline), T1 (1 week), T2 (1 month), T3 (6 months), T4 (12 months)
  MAAS means Mindful Attention Awareness Scale; this scale is a 15-item scale designed to assess a central characteristic of the state of mindfulness: an open or receptive awareness; higher scores reflect higher levels of dispositional mindfulness.The DASS-21 means Depression Anxiety and Stress Scale; this Scale assesses the emotional state: it is a clinical assessment lasting 3 minutes and 21 questions; It measures the three related states of depression, anxiety and stress; scores for depression, anxiety and stress are calculated by summing the scores for the relevant items.

CONTACTS AND LOCATIONS:
Overall Officials: Marlúcia S Jesus, Student, Principal Investigator — Federal University of São Paulo
Locations (1):
- Centro Mente Aberta em Mindfulness, São Paulo, Brazil

IPD SHARING:
Plan to Share IPD: Yes
Data will be shared by research gate.
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: December 2021. Will be available for 2 years
Access Criteria: Access will be granted to those researchers who are interested in developing studies with objectives similar to this research.

REFERENCES:
- [Background] Rothlin P, Birrer D, Horvath S, Grosse Holtforth M. Psychological skills training and a mindfulness-based intervention to enhance functional athletic performance: design of a randomized controlled trial using ambulatory assessment. BMC Psychol. 2016 Jul 26;4(1):39. doi: 10.1186/s40359-016-0147-y. PMID 27457721
- [Background] Buhlmayer L, Birrer D, Rothlin P, Faude O, Donath L. Effects of Mindfulness Practice on Performance-Relevant Parameters and Performance Outcomes in Sports: A Meta-Analytical Review. Sports Med. 2017 Nov;47(11):2309-2321. doi: 10.1007/s40279-017-0752-9. PMID 28664327
- [Background] Kozasa EH, Sato JR, Lacerda SS, Barreiros MA, Radvany J, Russell TA, Sanches LG, Mello LE, Amaro E Jr. Meditation training increases brain efficiency in an attention task. Neuroimage. 2012 Jan 2;59(1):745-9. doi: 10.1016/j.neuroimage.2011.06.088. Epub 2011 Jul 7. PMID 21763432
- [Background] Jones G. More than just a game: research developments and issues in competitive anxiety in sport. Br J Psychol. 1995 Nov;86 ( Pt 4):449-78. doi: 10.1111/j.2044-8295.1995.tb02565.x. PMID 8542197
- [Background] Hardy L, Jones G. Current issues and future directions for performance-related research in sport psychology. J Sports Sci. 1994 Feb;12(1):61-92. doi: 10.1080/02640419408732158. PMID 8158748
- [Background] Burns L, Weissensteiner JR, Cohen M. Lifestyles and mindsets of Olympic, Paralympic and world champions: is an integrated approach the key to elite performance? Br J Sports Med. 2019 Jul;53(13):818-824. doi: 10.1136/bjsports-2018-099217. Epub 2018 Oct 23. PMID 30352862
- [Background] Navarro-Haro MV, Lopez-Del-Hoyo Y, Campos D, Linehan MM, Hoffman HG, Garcia-Palacios A, Modrego-Alarcon M, Borao L, Garcia-Campayo J. Meditation experts try Virtual Reality Mindfulness: A pilot study evaluation of the feasibility and acceptability of Virtual Reality to facilitate mindfulness practice in people attending a Mindfulness conference. PLoS One. 2017 Nov 22;12(11):e0187777. doi: 10.1371/journal.pone.0187777. eCollection 2017. PMID 29166665
- [Background] Lutz A, Slagter HA, Dunne JD, Davidson RJ. Attention regulation and monitoring in meditation. Trends Cogn Sci. 2008 Apr;12(4):163-9. doi: 10.1016/j.tics.2008.01.005. Epub 2008 Mar 10. PMID 18329323
- See also: Conde, AJM. Memória Paralímpica. vol. I São Paulo: Comitê Paralímpico Brasileiro; 2018. Accessed June 15, 2019. — https://indd.adobe.com/view/0e47dd19-9663-4cd6-870e-072617bec30b?fbclid=IwAR3NY5enAgsrsEQcV93CZRAzsPCYF-UJaCvYTWbqMDjFZo3PUpwrohORtgU.
- See also: Winckler C, Oliveira MC. O esporte Paralímpico e os caminhos para a inclusão social. Revista Científica Virtual da ESA, v. 27, p. 176-186, 2018. Accessed June 15, 2019 — http://issuu.com/esa_oabsp/docs/revista_27_-_direito_desportivo
- See also: BISFed International Boccia Rules - 2018 (v.3). Accessed May 15, 2019. — http://www.bisfed.com/wp-content/uploads/2018/05/V.3_editable_boccia_rules-portuguese-BRA.pdf.
- See also: O que é Bocha. Accessed May 10, 2019. — http://ande.org.br/modalidades-bocha/
- See also: Kabat-Zinn J. Mindfulness-Based Interventions in Context: Past, Present, and Future. Clin Psychi-Sci Pract. 2003;10:144-56. Doi: 10.1093/clipsy.bpg0. — https://www.researchgate.net/publication/227546809_Mindfulness-Based_Interventions_in_Context_Past_Present_and_Future